CLINICAL TRIAL: NCT00745238
Title: Four Weeks Withdrawal of Non-invasive Ventilation (NIV) in Patients With Myotonic Dystrophy: Cardiovascular, Metabolic and Daytime Vigilance Induced Changes
Brief Title: Cardiovascular Consequences of NIV Withdrawal in Patients With Myotonic Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0801
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2008-09

CONDITIONS: Myotonia
Keywords: endothelial function; peripheral arterial tone; systemic inflammation; oxidative stress; respiratory and peripheral muscular function
MeSH Terms: conditions — Myotonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myotonic Dystrophy 1 (Experimental)
  Interventions: Other: withdrawal of non-invasive ventilation

INTERVENTIONS:
Other: withdrawal of non-invasive ventilation — Four weeks withdrawal of non-invasive ventilation

SUMMARY:
Background: Myotonic dystrophy lead to highly heterogeneous, multisystemic symptoms including myotonia, progressive muscle weakness, cardiac conduction defects, cataract, metabolic dysfunction, and excessive daytime somnolence. This last symptom is related to respiratory failure and/or to involvement of the central nervous system. However the metabolic disturbances could contribute to it. From the respiratory point of view this disease is characterised by the progressive appearance of respiratory failure of muscular origin but mainly associated with a defect in the central respiratory drive. The treatment for this hypoventilation is non-invasive ventilation (NIV).

It is not currently absolutely clear as to the best choice of criteria to judge long term effectiveness of NIV. The most usual criteria are normalisation of daytime blood gases, diminution of respiratory work, improvement in daytime symptoms and improvement in sleep structure. Other criteria are currently little studied, for instance the contribution of the interaction between alveolar hypoventilation and oxygen desaturation during the night and biological deficiencies such as systemic inflammation, glucose intolerance or insulin resistance. Likewise there is little information about the interaction between alveolar hypoventilation and endothelial dysfunction and arterial stiffness both being accurate predictive factors for cardiovascular risks.

Aim: to evaluate the impact of NIV on endothelial dysfunction in patients with myotonic dystrophy. The secondary objectives are to assess the impact of NIV on systemic inflammation, arterial stiffness, insulin-resistance, quality of sleep, and daytime vigilance in these patients.

Methods: Patients with chronic alveolar hypoventilation already treated by long term NIV will be included. They will have an initial check-up (Visit 1), then will interrupt NIV treatment for four weeks (Visit 2), and then return to NIV treatment. The last check-up will be done four weeks after NIV resumption (Visit3).

Expected results: It is expected that NIV withdrawal will results in a deterioration of cardio-vascular parameters (endothelial function and arterial stiffness), metabolic parameters (insulin-resistance and systemic inflammation), quality of sleep and daytime vigilance. Return to NIV treatment may show an improvement of these parameters with a basal state recovery.

DETAILED DESCRIPTION:
NIV is a technique of assisted ventilation that does not use the endotracheal route as the interface between the patient and the ventilator. NIV by positive pressure assistance involves ventilating the patient by means of a mask adjusted on the nose or covering the nose and mouth. This technique is now the recommended therapeutic strategy for the treatment of chronic alveolar hypoventilation. It improves survival and quality of life, and improves daytime blood gases in patients suffering form chronic restrictive respiratory failure.

For each check-up (3 visits), patients will have a polysomnography, a complete respiratory function measurement (Flows and lung volumes, CO2 sensitivity test, SNIF test, blood gazes analysis), a test of endothelial function (peripheral arterial tone), a test of arterial stiffness (pulse wave velocity), an assessment of systemic inflammation (ultra sensitive CRP, TNFa, IL6), assessment of diurnal vigilance tests ( OSLER test and sleepiness scale) and assessment of metabolic and endocrinal function (insulinemia, glucose blood level, Leptin, DHEA).

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients (>18 yrs) suffering from myotonic dystrophy already treated by long term nocturnal non invasive ventilation for more than six months for a chronic hypercapnic respiratory failure (Level of PaCO2 at beginning of the treatment should be between 45 and 55 mmHg)
* Patients should use his (her) non-invasive ventilation more than 4 hours and less than 12 hours per day.
* Patients could have an associated obstructive or/and central sleep apnea.
* NIV treatment should be consider as "efficient ": To allow an improvement of PaCO2 during wakefulness in the morning when using NIV compared to PaCO2 at the beginning of the treatment; To allow an improvement of the nocturnal oxymetry compared to baseline (mean nocturnal SaO2 > 90%).

EXCLUSION CRITERIA:

* Patients with a concomitant respiratory condition contributing to daytime alveolar hypoventilation.
* Patients judged by investigators as at high cardiovascular risk, this contraindicating NIV withdrawal.
* Patients with cardiac failure and periodic breathing.
* Patients who have had an acute episode of respiratory failure in the previous month.
* Incapacitated patients in accordance with article L 1121-6 of the public health code.
* Patients treated by oral corticosteroids or oral long-term non-steroidal anti-inflammatory drugs (NSAID).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate endothelial dysfunction (as measured by Peripheral arterial tone (PAT)) and its evolution after four weeks withdrawal of non-invasive ventilation (NIV). | 8 weeks

SECONDARY OUTCOMES:
To assess arterial stiffness, systemic inflammation (IL6, TNFα, Leptin, CRP), insulin resistance, DHEA, sleep quality, objective and subjective daytime somnolence and their evolution after four weeks withdrawal of NIV. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, PROFESSOR, Principal Investigator — University Hospital, Grenoble
Locations (1):
- France.Functional Cardio-Respiratory Exploration Laboratory, Grenoble, Isere, France

REFERENCES:
- [Background] 1-Cho DH. Biochim Biophys Acta 2007;1772:195-204. 2-Harper PS. W.B. Saunders ed. London, 1989. 3-Machuca-Tzili L. Muscle Nerve 2005;32:1-18. 4-Lazarus A. J Am Coll Cardiol 2002;40:1645-52. 5-Johansson A. J Intern Med 1999;245:345-51. 6-Johansson A. Int J Obes Relat Metab Disord 2002;26:1386-92. 7-Carter JN. J Clin Endocrinol Metab 1985;60:611-4. 8-Kouki T. Diabet Med 2005;22:346-7. 9-Mammarella. J Neurol Sci 2002;201:59-64. 10-Laberge L. J Sleep Res 2004;13:95-100. 11-Begin P. Am J Respir Crit Care Med 1997;156:133-9. 12-DAngelo MG. Muscle Nerve 2006;34:16-33. 13-Veale D. Eur Respir J 1995;8:815-8. 14-Vgontzas A. Sleep Med Rev 2005;9:211-24. 15-Perrin C. Semin Respir Crit Care Med 2005;26:117-30. 16-Guilleminault C. J Neurol Neurosurg Psychiatry 1998;65:225-32. 17-Mehta S. Am J Respir Crit Care Med 2001;163:540-77. 18-Babu AR. Arch Intern Med 2005;165(4):447-52. 19-Talbot K. Neuromuscul Disord 2003;13(5):357-64.